CLINICAL TRIAL: NCT05410301
Title: Feasibility Study of a Static Magnetic and Electric Field Device in Adults With Recurrent Glioblastoma and Their Partners
Brief Title: Golden Halo, Static Magnetic and Electric Field Device, in Recurrent Glioblastoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving institution
Sponsor: Varun Monga, MD (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor-Investigator, Varun Monga, MD, Clinical Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202109325
Record Dates: First submitted 2022-05-11; First posted 2022-06-08 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Glioblastoma; Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Lomustine; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Cohort 1 - Main study group consisting of patients with rGBM and Cohort 2 - Substudy group consisting of a participating unaffected partners of patients with rGBM
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Patients: sBE device applied during sleep, in combination with Lomustine and Bevacizumab (Experimental): The sBE device is to be used 8 hours a day by the patients, during sleep, for 8 weeks, while also receiving standard chemotherapy Lomustine and Bevacizumab
  Interventions: Device: Static Magnetic and Electric (sBE) device; Drug: Lomustine; Drug: Bevacizumab
- Partners of Patients (who sleep in same bed): sBE (Experimental): Up to 12 associated unaffected partners may agree to sleep within the investigational sBE device congruent with the period of exposure of their rGBM partner (8 weeks + possible extension)
  Interventions: Device: Static Magnetic and Electric (sBE) device

INTERVENTIONS:
Device: Static Magnetic and Electric (sBE) device — Home-based Static Magnetic and Electric (sBE) device that is slept in
Drug: Lomustine — Chemotherapy drug
  Arms: Patients: sBE device applied during sleep, in combination with Lomustine and Bevacizumab
Drug: Bevacizumab — Chemotherapy and targeted therapy drug
  Arms: Patients: sBE device applied during sleep, in combination with Lomustine and Bevacizumab

SUMMARY:
A prospective, open label, single-center, early feasibility trial will be conducted to assess the safety and feasibility of a home-based Static Magnetic and Electric (sBE) device applied for 8 hours/day during sleep in adult participants with recurrent glioblastoma (rGBM) at their first relapse.

DETAILED DESCRIPTION:
The purpose of this research study is to test the feasibility of a Static Magnetic and Electric Field (sBE) Device when combined with standard chemotherapy drugs, Lomustine and Bevacizumab, in the treatment of patients with recurrent glioblastoma.

The sBE device produces static magnetic (sB) and electric (sE) fields and is to be used 8 hours a day by the patients, during sleep, for 8 weeks, while also receiving standard chemotherapy Lomustine and Bevacizumab.

Patients will have visits in clinic every two weeks during the treatment period. The visits will include MRI scans, quality of life assessments, neurological and physical exams, and blood draws.

After the sBE treatment period, patients will continue standard chemotherapy with their regular oncologists.

Partners of the patients, who sleep in the same beds, will be invited to participate and will be involved in the study procedures except for those intended to monitor the disease. If partners do not agree to participate, they will not be able to sleep in the devices.

ELIGIBILITY:
Inclusion Criteria - Main Study Participants (Cohort 1) only

All participating subjects must meet the following criteria on the screening examination to be eligible to participate in the study:

* Participants must be able to understand and willing to sign a written informed consent document. The study requires authorization for collection, utilization and storage of biological materials (blood, plasma, serum) to be used for research on the effects of sBE on tissues.
* If the participant lives with a partner/spouse and they choose to participate in the study as part of Cohort 2, the partner/spouse must be able to understand and be willing to sign a written informed consent document. If the partner chooses not to participate they will be given specific instructions for sleeping arrangements and not being exposed to sBE therapy.
* Participants must allow the research team to assemble the sBE device in their homes and conduct in-person visits or video conference calls for technical support. Participants must reside within a 100 mile radius of Iowa City. Participants must participate in in-person training of use of the sBE device and understand how to safely use the sBE device, and agree to adhere to use only as instructed in the instruction manual (see Appendix I).
* Participants must be able to adhere to using the sBE device daily for at least 8 hours, adhere to the scheduled visits, and agree to record sBE device usage hours accurately and consistently in a daily diary.
* Participants must be 18 years of age or older on the day of signing the informed consent document.
* Participants must have a Karnofsky Performance Status (KPS) ≥ 60 (see Appendix B).
* Participants must be able to physically operate the sBE device independently or with the assistance of a caretaker (see Appendix I).
* Participants must allow a collection of blood/plasma during scheduled visits where labs will be collected for translational research study purposes.
* Participants must allow the study team to disassemble the sBE device and retrieve static magnetic and electric generating components at the termination of the study. Participants may keep the foam mattress or have it removed by the research team at the time of sBE device disassembly.
* Patients must have histologically confirmed GBM (primary) with unequivocal first progression of disease (confirmed by MRI or CT within 2 weeks of study registration).
* Patients must have previous history of failing temozolamide and radiation with this being the first recurrence after standard of care therapy.
* Patients must have no history of bleeding diathesis, previous intracranial hemmorhage, previous intolerance to lomustine or bevacizimab.
* If the patient has had surgical re-resection of the tumor, the following must be true:

  * The surgery must confirm the recurrence, but residual or measurable disease after surgery is not a requirement
  * An MRI must be taken within 48-96 hours following the surgery
  * Surgery must have been completed at least 2 weeks before starting treatment with the sBE device
* Patients must have recovered from acute sequelae of surgery. When use of the sBE device is initiated, the craniotomy or intracranial biopsy site must be adequately healed as determined by:

  * No drainage or cellulitis
  * No residual sutures or staples
  * Intact underlying cranioplasty (no craniectomy)
* Initiation of use with the sBE device must be > 2 weeks after the last tumor related surgical procedure.
* If the patient is taking steroids, the dose must be stable or decreasing for at least 5 days before the baseline scan and up to the start of the study therapy.
* Absence of any recent hemorrhagic or thrombotic events in the brain.

Clinical labs - must be performed within 14 business days prior to registration and determined to be within the reference ranges listed below:

* Hematology:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 109 cells/L
  * Platelet count ≥ 100 x 109 cells/L
  * Hemoglobin ≥ 9.9 g/dL
* Biochemistry:

  * Bilirubin < 1.5 x 1.2 mg/dL
  * AST < 2.5 x 40 U/L (males) and < 2.5 x 32 U/L (females)
  * ALT < 2.5 x 41 U/L (males) and < 2.5 x 33 U/L (females)
  * ALP < 2.5 x 129 U/L (males) and < 2.5 x 104 (females)
  * Plasma amylase ≤ 1.5 x 100 U/L
  * Plasma lipase ≤ 1.5 x 60 U/L
  * Creatinine < 1.5 x 1.2 mg/dL (males) and <1.5 x 1.0 mg/dL (females) or calculated 24 hour creatinine clearance ≥ 50 mL/min
  * Proteinuria (by urine dipstick) < 2. If ≥ 2 proteinuria on dipstick urinalysis at baseline, will need to undergo 24 hour urine collection and show ≤ 1 g protein within a 24 hour period.
  * Total plasma calcium (corrected for plasma albumin as needed) or ionized calcium within UIHC's reference range (8.6 - 10.3 mg/dL).
* Coagulation studies:

  * INR < 1.5
  * aPTT < 1.5 x 35 s, unless receiving therapeutic low molecular weight heparin
* Patients with a buffer range from the normal values of ± 5% for hematology and ± 10% for biochemistry are acceptable as determined by the investigator.

Pregnancy and Reproduction

* Women of child-bearing potential (WOCBP) must agree to use a medical contraceptive method during the treatment period and 6 months after the last dose of lomustine and bevacizumab or with sBE device use, whichever is later. WOCBP include any female who is not postmenopausal or has not undergone successful surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy). Women must not be breastfeeding. In general, appropriate methods of preventing pregnancy should be discussed and agreed upon by the investigator and study participant.

  * Acceptable contraception methods may include oral contraceptives, other hormonal contraceptives (implants, an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.
  * Post-menopause and not of child bearing potential is defined as 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with plasma FSH levels > 40 mIU/mL and estradiol < 20 pg/mL.
  * WOCBP must have a negative plasma or urine pregnancy test within 3 days prior to starting treatment with the sBE device.
* Men must agree to use a reliable method of birth control and to not donate sperm during the treatment period and for at least 6 months after the last dose of lomustine and bevacizumab or treatment with the sBE device, whichever is later.

Exclusion Criteria

Participants who meet any of the following criteria will not be eligible for admission into the study.

Previous Therapies

* Previous or current treatment with any investigational electromagnetic field generating devices, including but not limited to the Optune and Voyager devices.
* Definitive radiation therapy within three months before the diagnosis of disease progression. Palliative radiation 4 weeks prior to treatment is allowed.

Concomitant Medications & Devices

* Implanted electronic medical device including but not limited to implanted cardiac defibrillator, pacemaker, deep brain stimulator.
* Patients who take enzyme-inducing anti-epileptic drugs (EIAED) must be put on non-EIAED anti-convulsants at least 2 weeks prior to starting the lomustine and bevacizumab.
* Underlying conditions that may interfere with lomustine, bevacizumab, or the investigational sBE device within 6 months prior to study registration. If the medical investigator feels intercurrent illness (ie. Infection) prevents delivery of lomustine and bevacizumab they will be excluded.
* Current or recent use of anti-thrombotics or anti-coagulants including but not limited to the following criteria:

  * Use of aspirin > 325 mg/day or other NSAID with anti-platelet activity within 10 days of the first dose of bevacizumab
  * Treatment with dipyramidole, ticlopidine, clopidogrel, or cilostaz within 10 days of first dose of bevacizumab
  * Use of full dose anti-coagulants if patient's international normalized ratio (INR) > 1.5 x upper limit of the normal range (ULN) and activated prothrombin time (aPTT) > 1.5 x ULN. Use of full dose anti-coagulants is permissible if the INR or aPTT is within therapeutic limits according to the medical standards at UIHC and the patient is stable on the current dose for at least 14 days before starting investigational study.

Comorbidities

* History of known hypersensitivity to lomustine or bevacizumab formulations or chemical/biological similars, recombinant human antibodies, humanized antibodies, or Chinese hamster ovary cell products.
* Other previous malignancies, unless the patient was treated with curative intent > 2 years prior to registration and determined to be of low risk for recurrence as determined by the treating investigator, with the exception of well controlled basal cell carcinoma or squamous carcinoma of the skin or cervical cancer in situ.
* Hemorrhagic or thrombotic events within 6 months prior to study registration including but not limited to history or evidence of inherited bleeding or coagulation disorders, arterial or venous thromboses, history or evidence of stroke or TIAs, pulmonary embolisms, or pulmonary hemorrhage/hemoptysis greater than grade 1 according to the CTCAE v5.0 criteria within 1 month of study registration.
* Patients with any impairments in cardiac function within 6 months of the start of the study or clinically significant cardiac diseases, including but not limited to MI, severe/unstable angina, serious cardiac arrhythmias requiring medication or implanted devices (e.g. pacemaker or ICD), second/third degree heart block, history of or ongoing pericarditis, congestive heart failure (New York Heart Association functional classification III-IV), cardiomyopathy, congenital long QT syndrome, coronary artery bypass graft, aortic aneurysms requiring surgical intervention or peripheral arterial thromboses, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (defined by systolic BP > 150 mmHg and diastolic BP > 100 mmHg).
* Presence of an active or ongoing infection or serious underlying medical condition including but not limited to chronic liver disease, chronic kidney disease, chronic pulmonary disease, pancreatitis, or any other clinically relevant disease (other than GBM) that in the investigator's opinion would interfere with the study.
* Psychosocial illness or situations that would interfere with participant compliance to the study requirements.
* Any major systemic surgery ≤ 2 weeks prior to the initiation of the study.
* Patients who are pregnant or breastfeeding.
* Patients with a history of known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhage within 1 year of study registration.

SUBSTUDY PARTICIPANT SELECTION

The unaffected partner of the patient with recurrent GBM will be offered the option to participate in the substudy of the feasibility and safety of treatment with a sBE device. The unaffected partner must understand that their decision to participate or not participate in the substudy is completely voluntary and does not in any way impact the ability of their partner with rGBM to participate in the study. The same screening examination and evaluation will be conducted for the unaffected partner as the patient with recurrent GBM and are detailed in Section 10, Study Calendar. Within 2 weeks of registration, all assessments will occur unless otherwise noted. Each substudy participant must be fully informed on all aspects of the study for informed consent. If the unaffected partner wishes to participate in the substudy, the written informed consent must be obtained from the unaffected partner prior to enrollment of both the GBM patient and the unaffected partner.

Following registration, any additional laboratory assessments and/or start of medication that may alter tolerance to the prescribed combination of lomustine, bevacizumab and sBE may be used to re-assess eligibility.

Inclusion Criteria - Substudy Participants (Cohort 2) only

All substudy participants must meet the following criteria on the screening examination to be eligible to participate in the study:

* Able to understand and willing to sign a written informed consent document.
* Be the partner/spouse of a patient with rGBM and be cohabitating and sharing a bed with said patient with rGBM.
* Agree to allow the research team to assemble the sBE device in their homes and conduct in-person visits or video conference calls for technical support.
* Agree and be able to adhere to using the sBE device daily for at least 8 hours, adhere to the scheduled visits, and agree to record the number of hours using the sBE device accurately and consistently in a daily diary.
* Agree to getting a blood/plasma collection for translational research study purposes at scheduled visits where blood collections are outlined.
* Agree to accompany their partner with rGBM to all clinical visits where feasibility and safety assessments of the sBE device are being conducted.
* 18 years of age or older on the day of signing the informed consent document.
* Healthy as determined by screening assessment and the judgement of the principle investigator.
* Able to physically operate the sBE device according to the provided instruction manual (see Appendix I).
* Willing to end treatment with the sBE device when their partner with rGBM terminates treatment with the sBE device.
* Willing to allow the study team to disassemble and retrieve the static magnetic and electric generating components of the sBE device at the termination of the study.
* WOCBP must agree to use a medical contraceptive method during the 2-month period of using the sBE device and 6 months after the treatment with the sBE device. WOCBP include any female who is not postmenopausal or has not undergone successful surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy). Women must not be breastfeeding. In general, appropriate methods of preventing pregnancy should be discussed and agreed upon by the investigator and study participant.
* Acceptable contraception methods may include oral contraceptives, other hormonal contraceptives (implants, an intrauterine device [IUD] or barrier method. If condoms are used as a barrier method, a spermicidal agent should be added as a double barrier protection.

  * Post-menopause and not of child bearing potential is defined as 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with plasma FSH levels > 40 mIU/mL and estradiol < 20 pg/mL.
  * WOCBP must have a negative plasma or urine pregnancy test within 3 days prior to starting treatment with the sBE device.
* Men must agree to use a reliable method of birth control and to not donate sperm during the treatment period and for at least 6 months after treatment with the sBE device.

Exclusion Criteria

* Clinically relevant history or current presence of severe comorbidities as determined by the principle investigator including but not limited to cardiovascular, neurological, respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, or psychiatric diseases.
* Previous malignancies, unless the participant was treated with curative intent >2 years prior to registration or determined to be of low risk for recurrence by the primary investigator, with the exception of well controlled basal cell carcinoma or squamous carcinoma of the skin or cervical cancer in situ.
* Implanted electronic medical device including but not limited to implanted cardiac defibrillator, pacemaker, deep brain stimulator
* Current or recent (within 4 weeks of before starting use of the sBE device) treatment with any investigational drug(s) or device(s).
* History of seizures or current use of enzyme-inducing anti-epileptic drugs (EIAED).
* Any impairments in cardiac function within 6 months of the start of the study or clinically significant cardiac diseases including but not limited to MI, severe/unstable angina, serious cardiac arrhythmias requiring medication or implanted devices (e.g. pacemaker or ICD), second/third degree heart block, history of or ongoing pericarditis, congestive heart failure (New York Heart Association functional classification III-IV), cardiomyopathy, congenital long QT syndrome, coronary artery bypass graft, aortic aneurysms requiring surgical intervention or peripheral arterial thromboses, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (defined by systolic BP > 150 mmHg and diastolic BP > 100 mmHg).
* Presence of an active or ongoing infection or serious underlying medical condition including but not limited to chronic liver disease, chronic kidney disease, chronic pulmonary disease, pancreatitis, or any other clinically relevant disease that in the investigator's opinion would interfere with the study.
* Psychosocial illness or situations that would interfere with participant compliance to the study requirements.
* Any major systemic surgery ≤2 weeks prior to the initiation of the study.
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Greater than or equal to 80% sBE compliance as determined by device pressor sensors, participant reporting via daily diary, and participant completion of sBE Device Questionnaire | From initiation of therapy through 8 weeks of therapy
  sBE device use will be assessed based on participant compliance. Compliance will be assessed using sensors in the sBE device, self-reporting via a daily diary, and the sBE Device Questionnaire administered approximately every 2 weeks during the initial 8-week sBE administration period (to coincide with a cycle of lomustine or bevacizumab for Cohort 1 participants).
Adverse Events according to CTCAE v5.0 | During the initial 8 weeks of treatment
  Safety of daily treatment with sBE as determined by the absence of Grade 3 adverse events attributable to sBE as outlined by the CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Varun Monga, MD, Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No